CLINICAL TRIAL: NCT04225403
Title: Telephone-based Motivational Interviewing Delivered by IBD ( Inflammatory Bowel Disease) Nurses for Smoking Cessation in Crohn's Disease: a Randomized Open-label Clinical Trial
Brief Title: Telephone-based Motivational Interviewing for Smoking Cessation in Crohn's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: GETTEII ( Grupo Enfermero de Trabajo en Enfermedad Inflamatoria Intestinal (Unknown); Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PR(AG)275/2013
Record Dates: First submitted 2019-12-23; First posted 2020-01-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Crohn Disease
Keywords: Inflammatory Bowel Disease; Smoking cessation; Tobacco; Smoking; Advanced practice nurse; Motivational intervention
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Smoking Cessation; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone-based motivational interviewing (Experimental): Experimental intervention consisted of a motivational intervention for smoking cessation through telephone every 3 months for one year, performed by IBD nurse
  Interventions: Behavioral: Telephone-based motivational interviewing for smoking cessation
- usual care (No Intervention): No intervention consisted of a single telephone contact one year after the star of the study

INTERVENTIONS:
Behavioral: Telephone-based motivational interviewing for smoking cessation — The motivational brief intervention is known by the acronym 5 R and lasts about 5-10 minutes. It is an approach based on the principles of motivational interviewing and develops the intervention in five short steps:
  * Relevance. Help patients identify why personal reasons may be relevant to quitting smoking.
  * Risks. Help identify what negative consequences tobacco use has.
  * Rewards. Help identify potential benefits of quitting smoking.
  * Resistors. Help patients identify barriers to smoking cessation, which can often include fear of withdrawal symptoms, failure, wainweight, face social situations, etc.
  * Repeat. Repeat the intervention at 3 months if you do not advance at the stage of change.
  Arms: Telephone-based motivational interviewing

SUMMARY:
Quitting smoking unequivocally improves the course of Crohn's disease (EC), and therefore, it should be one of the main therapeutic targets in the treatment of this disease. The goal of the study was to know the effectiveness of motivational intervention 5 R for smoking cessation in patients with Crohn's disease performed by telephone by nursing, in relation to those who did not receive such intervention.

For this purpose, a controlled, randomized, parallel and open clinical trial was designed. The subjects were patients with Crohn's disease that were actively smoking EC. They were all >18 years old and they had internet access and e-mail. Those who were already in a process of smoking cessation were excluded from the study. Experimental intervention consisted of a motivational intervention for smoking cessation through telephone every 3 months for one year.

ELIGIBILITY:
Inclusion Criteria:

* Smokers Crohn's disease patients
* >18 age

Exclusion Criteria:

* Smokers Crohn's disease patients who are receiving treatment of tobacco cessation at the time of inclusion
* Do not have email

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Change from motivation to quit smoking after at one year in the control group and in the experimental group | We measure it at baseline and through study completion, 1 year after
  Test de Richmond: to measure the motivation to quit smoking. It consists of 4 questions, scores from 0 to 10, highest score, highest motivation. It provides three categories, low motivation <4 points, medium motivation 5-6 and high motivation ≥7
Change from stages of changes to quit smoking after at one year in the control group and in the experimental group | We measure it at baseline and through study completion, 1 year after
  Stages of changes form Prochaska / DiClemente. Transtheoretical model of change consists of 4 mutually exclusive questions and has a legend where it classifies patients according to the state of the wheel of change in which they are: pre-contemplation, preparation, action, maintenance, consolidation and relapse.

SECONDARY OUTCOMES:
Number of patients with Crohn's disease who quit smoking at the end of the study in the control group and in the experimental group. | We measure it at baseline and through study completion, 1 year after
  Cosnes classification: current smokers >7 cigarettes per week for at least 6 months, former smokers who had stopped smoking at least 6 months before.

OTHER OUTCOMES:
The rate of patients who had received the 5 A intervention referred to the smoking cessation unit. | We measure it at baseline and through study completion, 1 year after
  Control visits in Hospital smoking cessation Unit
The rate of patients who had received the 5 R intervention referred to the smoking cessation unit. | We measure it at baseline and through study completion, 1 year after
  Control visits in Hospital smoking cessation Unit

CONTACTS AND LOCATIONS:
Overall Officials: Ester Navarro Correal, MsC, Principal Investigator — Hospital Universitari Vall d'Hebron Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cosnes J, Beaugerie L, Carbonnel F, Gendre JP. Smoking cessation and the course of Crohn's disease: an intervention study. Gastroenterology. 2001 Apr;120(5):1093-9. doi: 10.1053/gast.2001.23231. PMID 11266373
- [Result] Kaplan GG. Smoking Cessation for Crohn's Disease: Clearing the Haze. Am J Gastroenterol. 2016 Mar;111(3):420-2. doi: 10.1038/ajg.2016.45. PMID 27018116
- [Result] Kemp K, Dibley L, Chauhan U, Greveson K, Jaghult S, Ashton K, Buckton S, Duncan J, Hartmann P, Ipenburg N, Moortgat L, Theeuwen R, Verwey M, Younge L, Sturm A, Bager P. Second N-ECCO Consensus Statements on the European Nursing Roles in Caring for Patients with Crohn's Disease or Ulcerative Colitis. J Crohns Colitis. 2018 Jun 28;12(7):760-776. doi: 10.1093/ecco-jcc/jjy020. No abstract available. PMID 29509882
- [Result] Underner M, Perriot J, Cosnes J, Beau P, Peiffer G, Meurice JC. [Smoking, smoking cessation and Crohn's disease]. Presse Med. 2016 Apr;45(4 Pt 1):390-402. doi: 10.1016/j.lpm.2016.02.008. Epub 2016 Mar 23. French. PMID 27016849
- [Result] Cosnes J. Smoking and Diet: Impact on Disease Course? Dig Dis. 2016;34(1-2):72-7. doi: 10.1159/000442930. Epub 2016 Mar 16. PMID 26981632
- [Result] To N, Gracie DJ, Ford AC. The Importance of Smoking Cessation in Improving Disease Course in Crohn's Disease. Am J Gastroenterol. 2016 Aug;111(8):1198. doi: 10.1038/ajg.2016.165. No abstract available. PMID 27481416
- [Derived] Navarro Correal E, Casellas Jorda F, Borruel Sainz N, Robles Alonso V, Herrera de Guise C, Ibarz Casas A, Sanchez Garcia JM, Vila Morte G, Fuentelsaz Gallego C. Effectiveness of a Telephone-Based Motivational Intervention for Smoking Cessation in Patients With Crohn Disease: A Randomized, Open-Label, Controlled Clinical Trial. Gastroenterol Nurs. 2021 Nov-Dec 01;44(6):418-425. doi: 10.1097/SGA.0000000000000572. PMID 34269705